CLINICAL TRIAL: NCT00004287
Title: Phase I Study of the Third Generation Adenovirus H5.001CBCFTR in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Pennsylvania (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11715; UPHS-28051
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases

INTERVENTIONS:
Genetic: H5.001CBCFTR

SUMMARY:
OBJECTIVES:

I. Assess the safety and feasibility of gene transfer with the third generation adenovirus H5.001CBCFTR in patients with cystic fibrosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: H5.001CBCFTR, an adenovirus vector containing the cystic fibrosis transmembrane conductance regulator gene, is administered endobronchially.

Cohort of 2 patients receive 1 of 6 H5.001CBCFTR concentrations. There is no intrapatient dose escalation.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Cystic fibrosis diagnosed as follows: Sweat sodium or chloride greater than 60 mEq/L by pilocarpine iontophoresis or cystic fibrosis genotype Clinical manifestations Estimated 2-year survival greater than 50%, i.e.: FEV1 at least 30% of predicted PaO2 greater than 55 mm Hg on room air PaCO2 less than 50 mm Hg on room air --Prior/Concurrent Therapy-- At least 2 months since systemic glucocorticoids At least 90 days since participation in investigational therapeutic study --Patient Characteristics-- Pulmonary: No pneumothorax within 12 months No asthma or allergic bronchopulmonary aspergillosis requiring glucocorticoids within 2 months No sputum pathogens unless sensitive to at least 2 antibiotics No hemoptysis of more than 250 mL blood over 24 hours within 1 year Other: No active adenoviral infection Ad5 (or similar type) antibody seropositive No other contraindication to protocol participation, e.g.: Drug abuse Alcoholism Psychiatric instability Inadequate motivation Documented azoospermia (men) Bilateral tubal ligation or hysterectomy (women) Screening exams within 4 weeks prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 1995-11

CONTACTS AND LOCATIONS:
Overall Officials: James M. Wilson, Study Chair — University of Pennsylvania

REFERENCES:
- [Background] Zuckerman JB, Robinson CB, McCoy KS, Shell R, Sferra TJ, Chirmule N, Magosin SA, Propert KJ, Brown-Parr EC, Hughes JV, Tazelaar J, Baker C, Goldman MJ, Wilson JM. A phase I study of adenovirus-mediated transfer of the human cystic fibrosis transmembrane conductance regulator gene to a lung segment of individuals with cystic fibrosis. Hum Gene Ther. 1999 Dec 10;10(18):2973-85. doi: 10.1089/10430349950016384. PMID 10609658